CLINICAL TRIAL: NCT04405856
Title: Outcome of Patients Treated With Intra Aortic Balloon Pump
Brief Title: Outcome of Patients Treated With IABP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Department of Cardiac Surgery, Nanjing Medical University
Other Study IDs: IABP-Jsph
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Acute Coronary Syndrome; Cardiogenic Shock; Coronary Artery Disease; Heart Failure; Left Ventricular Dysfunction; Low Cardiac Output Syndrome; Post-cardiac Surgery
MeSH Terms: conditions — Acute Coronary Syndrome; Shock, Cardiogenic; Coronary Artery Disease; Heart Failure; Ventricular Dysfunction, Left; Cardiac Output, Low | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intra Aortic Balloon Pump — Intra Aortic Balloon Pump (IABP) is a circulatory mechanical support device, placed in descending aorta, distally from left subclavian artery and proximally from renal artery. IABP works with counterpulsation concept, synchronized with heart cycle.

SUMMARY:
Intra-Aortic Balloon Pumps (IABP) is a widely used and effective left ventricular adjuvant therapy. IABP is an inflatable device placed in the aorta that inflates with diastole and deflates with systole. The aim of this study is to investigate the outcome of patients treated With IABP, and to evaluate the short-term and long-term outcomes of patients with IABP.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving IABP for circulatory support

Exclusion Criteria:

* Refusal of consent

Ages: 1 Year to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving IABP for circulatory support
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 30 days after IABP implantation

SECONDARY OUTCOMES:
All-cause mortality | 3 months after IABP implantation

CONTACTS AND LOCATIONS:
Overall Officials: Yong-feng Shao, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided